CLINICAL TRIAL: NCT02091375
Title: A Double Blind, Placebo Controlled Two-part Study to Investigate the Dose-ranging Safety and Pharmacokinetics, Followed by the Efficacy and Safety of Cannabidiol (GWP42003-P) in Children and Young Adults With Dravet Syndrome
Brief Title: Antiepileptic Efficacy Study of GWP42003-P in Children and Young Adults With Dravet Syndrome (GWPCARE1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP1332 Part B; 2014-002941-23 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy; Dravet Syndrome
Keywords: Cannabidiol; CBD; Epidiolex; GWP42003-P
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GWP42003-P 20 mg/kg/day Dose (Experimental): Participants received 20 mg/kg/day of GWP42003-P administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 20 mg/kg/day over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day) period.
  Interventions: Drug: GWP42003-P 20 mg/kg/day Dose
- Placebo (Placebo Comparator): Participants received placebo (0 mg/mL CBD), volume-matched to the 20 mg/kg/day dose level, administered orally, half in the morning and half in the evening. To maintain the blinded aspect of the study, participants titrated the placebo dose over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day of the matched dose) period.
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: GWP42003-P 20 mg/kg/day Dose — GWP42003-P was an oral solution containing 100 mg/milliliter (mL) cannabidiol (CBD) dissolved in the excipients, sesame oil and anhydrous ethanol (79 mg/mL), with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL).
  Other Names: Cannabidiol; Epidiolex
  Arms: GWP42003-P 20 mg/kg/day Dose
Drug: Placebo control — Placebo oral solution contained the excipients, sesame oil and anhydrous ethanol (79 mg/mL), with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL).
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To investigate the potential antiepileptic effects of cannabidiol (GWP42003-P) in children and young adults with Dravet syndrome.

DETAILED DESCRIPTION:
GWEP1332 Part B recruited an entirely new group of participants than GWEP1332 Part A. Participants who failed the entry criteria for Part A were eligible to take part in Part B.

Part B was a 1:1 randomized, double-blind, placebo-controlled, 14-week comparison of GWP42003-P versus placebo. The aim of Part B was to assess the antiepileptic efficacy of GWP42003-P as an adjunctive antiepileptic treatment compared with placebo, with respect to the percentage change from baseline during the treatment period of the study in convulsive seizure frequency in children and young adults.

Following the establishment of initial eligibility and baseline measurements, participants entered Part B and began a 28-day baseline observation period.

Eligible participants were then randomized to receive either GWP42003-P or placebo on a 1:1 basis and titrated up to the target dose that was identified in Part A (up to 20 milligrams [mg] per kilogram [kg] per day), which was confirmed following completion of Part A by an independent Data Safety Monitoring Committee who reviewed unblinded safety and pharmacokinetic data from Part A.

Participants received investigational medicinal product for 14 weeks, consisting of a titration period followed by a 12-week maintenance period.

Efficacy and safety were monitored at various clinic visits and via telephone. After 14 weeks of treatment, all participants were offered the option of entering an open label extension (OLE) study. Entry was within seven days of the final treatment visit. Participants who did not immediately enter the OLE study commenced a down-titration taper period lasting up to 10 days. The taper period was interrupted if the participant wished to enter the open label extension study within the seven-day timeframe.

For participants who opted not to enter the OLE study, a follow-up telephone call was made 28 days after the end of dosing and weekly safety telephone calls were made during the 28-day follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants were male or female aged between 2 and 18 years (inclusive).
* Participants had a documented history of Dravet Syndrome that was not completely controlled by current antiepileptic drugs.
* Participants took one or more antiepileptic drugs at a dose that had been stable for at least four weeks.
* All medications or interventions for epilepsy (including ketogenic diet and vagus nerve stimulation) were stable for four weeks prior to screening and participants were willing to maintain a stable regimen throughout the study.

Key Exclusion Criteria:

* Participants had clinically significant unstable medical conditions other than epilepsy.
* Participants had clinically relevant symptoms or a clinically significant illness in the four weeks prior to screening or randomization, other than epilepsy.
* Participants were currently using or had in the past used recreational or medicinal cannabis or synthetic cannabinoid based medications (including Sativex®) within the three months prior to study entry and were unwilling to abstain for the duration for the study.
* Participants had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal products.
* Participants had been part of a previous clinical trial involving another investigational product in the previous six months.
* There were plans for the participants to travel outside their country of residence during the study.
* Participants previously randomized into this study. In particular, participants who participated in Part A of the study could not enter Part B.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2015-11-26 (Actual); Study Completion 2015-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (13):
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Boston, Massachusetts
  - Rochester, Minnesota
  - New York, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Salt Lake City, Utah
- France (4):
  - Marseille
  - Paris
  - Strasbourg
  - Toulouse
- Poland (2):
  - Gdansk
  - Krakow
- United Kingdom (3):
  - Glasgow
  - Liverpool
  - London

REFERENCES:
- [Background] Devinsky O, Cross JH, Laux L, Marsh E, Miller I, Nabbout R, Scheffer IE, Thiele EA, Wright S; Cannabidiol in Dravet Syndrome Study Group. Trial of Cannabidiol for Drug-Resistant Seizures in the Dravet Syndrome. N Engl J Med. 2017 May 25;376(21):2011-2020. doi: 10.1056/NEJMoa1611618. PMID 28538134
- [Derived] Madan Cohen J, Checketts D, Dunayevich E, Gunning B, Hyslop A, Madhavan D, Villanueva V, Zolnowska M, Zuberi SM. Time to onset of cannabidiol treatment effects in Dravet syndrome: Analysis from two randomized controlled trials. Epilepsia. 2021 Sep;62(9):2218-2227. doi: 10.1111/epi.16974. Epub 2021 Jul 15. PMID 34265088

RESULTS

PARTICIPANT FLOW:
Groups:
- GWP42003-P 20 mg/kg/Day Dose: Participants received 20 milligrams (mg) per kilogram (kg) per day of GWP42003-P administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 20 mg/kg/day over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the open-label extension (OLE) study, the maintenance period was followed by a 10-day taper (10% per day) period.
- Placebo: Participants received placebo (0 mg/mL cannabidiol [CBD]), volume-matched to the 20 mg/kg/day dose level, administered orally, half in the morning and half in the evening. To maintain the blinded aspect of the study, participants titrated the placebo dose over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day of the matched dose) period.
Period: Overall Study
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Started | 61 | 59
Safety Analysis Set (All randomized participants who received at least 1 dose of investigational medicinal product (IMP)) | 61 | 59
Intention to Treat (ITT) Analysis Set (All participants in the Part B Safety Analysis Set who had post-baseline efficacy data) | 61 | 59
Completed | 52 | 56
Not Completed | 9 | 3
Not completed — Adverse Event | 8 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Withdrawn by the investigator | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: included all participants randomized to treatment who received at least 1 dose of IMP. Participants were analyzed according to the actual treatment they received.
Groups:
- GWP42003-P 20 mg/kg/Day Dose: Participants received 20 mg/kg/day of GWP42003-P administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 20 mg/kg/day over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day) period. Participants received at least 1 dose of IMP; analyzed according to the actual treatment received (GWP42003-P).
- Placebo: Participants received placebo (0 mg/mL CBD), volume-matched to the 20 mg/kg/day dose level, administered orally, half in the morning and half in the evening. To maintain the blinded aspect of the study, participants titrated the placebo dose over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day of the matched dose) period. Participants received at least 1 dose of IMP; analyzed according to the actual treatment received (placebo).
- Total: Total of all reporting groups
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.736 (4.7309) | 9.779 (4.8505) | 9.757 (4.7699)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 35 | 27 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline In Convulsive Seizure Frequency During The Treatment Period
Description: Convulsive seizures (atonic, clonic, tonic, or tonic-clonic) were recorded by the participant or caregiver using an interactive voice response system (IVRS) diary. Percentage change from baseline was calculated as: ([frequency during the treatment period - frequency during baseline]/frequency during baseline) * 100. The frequency during each period was based on 28-day averages and calculated as: (number of seizures in the period/number of reported days in the IVRS period) * 28. Baseline included all available data prior to Day 1 (28-day average). Negative percentages show an improvement from baseline.
Time Frame: Baseline to End of Treatment (EOT) (Day 99) or Early Termination (ET)
Population: ITT analysis set: included all participants in the Part B safety analysis set who had post-baseline efficacy data. Participants were analyzed according to the treatment group to which they were randomized. The ITT analysis set was the primary analysis set for all efficacy outcome measures.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 61 | 59
percent change | -38.94 [-69.53 to -4.83] | -13.29 [-52.53 to 20.20]
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0123, Wilcoxon rank-sum test; Median Difference (Final Values) = -22.79, 95% CI 2-sided [-41.06 to -5.43] — Calculated using the Hodges-Lehmann approach

2. Secondary Outcome: Number Of Participants With A ≥50% Reduction From Baseline In Convulsive Seizure Frequency During The Treatment Period
Description: Convulsive seizures (atonic, clonic, tonic, or tonic-clonic) were recorded by the participant or caregiver using an IVRS diary. Percentage change from baseline was calculated as per the primary outcome measure.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 61 | 59
Participants | 26 | 16
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0784, Cochran-Mantel-Haenszel; Stratified by age group (2-5 years, 6-12 years, and 13-18 years); Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.93 to 4.30]

3. Secondary Outcome: Number of Participants With A ≥25%, ≥75% Or 100% Reduction From Baseline In Convulsive Seizure Frequency During The Treatment Period
Description: as for outcome 2
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 61 | 59
Participants
  ≥25% Reduction | 38 | 26
  ≥75% Reduction | 14 | 7
  100% Reduction | 3 | 0

4. Secondary Outcome: Percentage Change From Baseline In Non-Convulsive Seizure Frequency During The Treatment Period
Description: Non-convulsive seizures (myoclonic, partial, or absence) were recorded by the participant or caregiver using an IVRS diary. Percentage change from baseline was calculated as per the primary outcome measure. Only participants with non-convulsive seizures during the baseline period were included. Negative percentages show an improvement from baseline.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 37 | 41
percent change | -40.16 [-92.1 to -3.6] | -34.69 [-97.5 to -0.7]

5. Secondary Outcome: Caregiver Global Impression Of Change In Seizure Duration (CGICSD)
Description: Seizure duration was assessed qualitatively using the CGICSD. Caregivers were asked "Since the patient started treatment, please assess the average duration of the patient's seizures (comparing their condition now to their condition before treatment)"; responses included decrease, no change, or increase in average duration. For each seizure type, only participants with at least 1 seizure for the corresponding seizure type, reported at any time during the study, were included.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 61 | 59
Participants
  Tonic-Clonic Seizures: number analyzed (Participants) | 49 | 41
  Tonic-Clonic Seizures: Decrease in average duration | 17 | 8
  Tonic-Clonic Seizures: No change in average duration | 32 | 31
  Tonic-Clonic Seizures: Increase in average duration | 0 | 2
  Tonic Seizures: number analyzed (Participants) | 12 | 15
  Tonic Seizures: Decrease in average duration | 4 | 2
  Tonic Seizures: No change in average duration | 8 | 12
  Tonic Seizures: Increase in average duration | 0 | 1
  Clonic Seizures: number analyzed (Participants) | 11 | 7
  Clonic Seizures: Decrease in average duration | 5 | 3
  Clonic Seizures: No change in average duration | 6 | 3
  Clonic Seizures: Increase in average duration | 0 | 1
  Atonic Seizures: number analyzed (Participants) | 3 | 7
  Atonic Seizures: Decrease in average duration | 2 | 2
  Atonic Seizures: No change in average duration | 1 | 3
  Atonic Seizures: Increase in average duration | 0 | 2
  Myoclonic Seizures: number analyzed (Participants) | 14 | 18
  Myoclonic Seizures: Decrease in average duration | 4 | 3
  Myoclonic Seizures: No change in average duration | 10 | 12
  Myoclonic Seizures: Increase in average duration | 0 | 3
  Countable Partial Seizures: number analyzed (Participants) | 12 | 13
  Countable Partial Seizures: Decrease in average duration | 5 | 2
  Countable Partial Seizures: No change in average duration | 7 | 9
  Countable Partial Seizures: Increase in average duration | 0 | 2
  Other Partial Seizures: number analyzed (Participants) | 3 | 5
  Other Partial Seizures: Decrease in average duration | 0 | 3
  Other Partial Seizures: No change in average duration | 3 | 2
  Other Partial Seizures: Increase in average duration | 0 | 0
  Absence Seizures: number analyzed (Participants) | 16 | 19
  Absence Seizures: Decrease in average duration | 4 | 6
  Absence Seizures: No change in average duration | 11 | 12
  Absence Seizures: Increase in average duration | 1 | 1

6. Secondary Outcome: Number Of Participants Using Rescue Medication
Description: The use of rescue medication was recorded by the participant or caregiver using a paper diary.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 61 | 59
Participants | 36 | 41

7. Secondary Outcome: Number Of Participants With Inpatient Hospitalizations Due To Epilepsy
Description: Inpatient hospitalizations due to epilepsy were recorded by the participant or caregiver and through the serious adverse events (SAE) reporting process.
Time Frame: Baseline to Safety Follow-up (Day 137)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 61 | 59
participants
  Caregiver/participant-reported | 5 | 1
  Investigator-reported (serious TEAE) | 2 | 1

8. Secondary Outcome: Change From Baseline In Sleep Disruption 0 To 10 Numerical Rating Scale (0 to 10 NRS) Score
Description: The sleep disruption 0 to 10 NRS questionnaire was completed by the participant's caregiver. The caregiver was asked 'On a scale of '0 to 10', please indicate the number that best describes your child's sleep disruption in the last week.' The markers ranged from 0 = 'slept extremely well' to 10 = 'unable to sleep at all'. The change from baseline in the sleep disruption 0 to 10 numerical rating scale score was analyzed using an analysis of covariance (ANCOVA) model with baseline and age group (2 to 5 years, 6 to 12 years and 13 to 18 years) as covariates and treatment group as a fixed factor. A negative change from baseline represents an improvement in sleep. Last visit for endpoints assessed at clinic visits was defined as the last scheduled visit (not including the end of taper or safety follow-up visits) at which participant's last evaluation was performed.
Time Frame: Baseline to Last Visit (Day 99) or ET
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 59 | 59
units on a scale | -0.7 [-1.5 to 0.1] | -0.3 [-1.1 to 0.5]

9. Secondary Outcome: Change From Baseline In Epworth Sleepiness Scale (ESS) Score
Description: The ESS questionnaire was completed by the participant's caregiver. The change from baseline in the ESS score was analyzed using an ANCOVA model with baseline and age group (2 to 5 years, 6- to 2 years and 13 to 18 years) as covariates and treatment group as a fixed factor. The total score was the sum of the 8 item-scores and ranged from 0 to 24. A higher total score represents greater levels of daytime sleepiness.
Time Frame: Baseline to Last Visit (Day 99) or ET
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 61 | 58
units on a scale | 0.82 [-0.36 to 1.99] | -0.69 [-1.90 to 0.52]

10. Secondary Outcome: Change From Baseline In Quality Of Life In Childhood Epilepsy (QOLCE) Score
Description: The QOLCE questionnaire was completed by the parent or caregiver of participants aged 4 years and above. The change from baseline in the overall quality of life score was analyzed using an ANCOVA model with baseline and age group (2 to 5 years, 6 to 12 years and 13 to 18 years) as covariates and treatment group as a fixed factor. Zero represents the lowest or poorest category and 100 represents the highest level of functioning. The overall quality of life score was calculated by taking the mean of the subscale scores.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 47 | 44
units on a scale | 5.6 [1.9 to 9.3] | 4.1 [0.2 to 8.0]

11. Secondary Outcome: Change From Baseline In Vineland Adaptive Behavior Scales, Second Edition (Vineland-II) Score
Description: The Vineland-II scores (standard scores and adaptive levels for each adaptive behavior domain, the adaptive behavior composite, and the maladaptive behavior index score and level) were assessed by the participant's caregiver. Scores were analyzed using an ANCOVA model with baseline and age group (2 to 5 years, 6 to 12 years, and 13 to 18 years) as covariates and treatment group as a fixed factor. Higher scores represent greater levels of functioning except for the maladaptive behavior index, for which a negative change from baseline represents an improvement in condition.
Time Frame: Baseline to Last Visit (Day 99) or ET
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 61 | 59
units on a scale
  Communication Domain Standard Score: number analyzed (Participants) | 17 | 19
  Communication Domain Standard Score | -0.8 [-3.2 to 1.5] | 3.0 [0.8 to 5.3]
  Daily Living Skills Domain Standard Score: number analyzed (Participants) | 20 | 19
  Daily Living Skills Domain Standard Score | -0.8 [-4.0 to 2.4] | -0.8 [-4.1 to 2.6]
  Socialization Domain Standard Score: number analyzed (Participants) | 12 | 16
  Socialization Domain Standard Score | -0.6 [-4.6 to 3.5] | -0.6 [-4.0 to 2.7]
  Motor Skills Domain Standard Score: number analyzed (Participants) | 20 | 22
  Motor Skills Domain Standard Score | -2.5 [-5.5 to 0.5] | 1.7 [-1.1 to 4.5]
  Adaptive Behavior Composite Standard Score: number analyzed (Participants) | 12 | 15
  Adaptive Behavior Composite Standard Score | -2.0 [-5.2 to 1.1] | 0.6 [-2.1 to 3.3]
  Maladaptive Behavior Index v-Scale Score: number analyzed (Participants) | 47 | 48
  Maladaptive Behavior Index v-Scale Score | -0.3 [-0.7 to 0.1] | -0.4 [-0.8 to 0.0]

12. Secondary Outcome: Caregiver Global Impression Of Change (CGIC)
Description: The CGIC was used to assess the participant's overall condition on a 7-point scale using the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse, or very much worse" (1 = very much improved; 7 = very much worse). On Day 1 (prior to starting IMP), the caregiver was asked to write a brief description of the participant's overall condition as a memory aid for the CGIC questionnaire at subsequent visits.
Time Frame: Baseline to Last Visit (Day 99) or ET
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 60 | 58
Participants
  Very Much Improved | 9 | 4
  Much Improved | 10 | 4
  Slightly Improved | 18 | 12
  No Change | 15 | 31
  Slightly Worse | 3 | 6
  Much Worse | 4 | 1
  Very Much Worse | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) to Day 137
Description: Included all participants randomized to treatment who received at least 1 dose of IMP. Participants were analyzed according to the actual treatment they received.
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 10/61 | 3/59
Other Adverse Events (participants affected / at risk) | 46/61 | 28/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 20 mg/kg/Day Dose (N=61) | Placebo (N=59)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Platelet count (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 3 | 3
Convulsion (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 3 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 20 mg/kg/Day Dose (N=61) | Placebo (N=59)
Diarrhoea (Gastrointestinal disorders) | 19 | 6
Vomiting (Gastrointestinal disorders) | 9 | 3
Pyrexia (General disorders) | 9 | 5
Fatigue (General disorders) | 11 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Nasopharyngitis (Infections and infestations) | 3 | 3
Gamma-glutamyltransferase increased (Investigations) | 4 | 0
Transaminases increased (Investigations) | 4 | 0
Weight decreased (Investigations) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 16 | 3
Somnolence (Nervous system disorders) | 19 | 6
Lethargy (Nervous system disorders) | 7 | 3
Headache (Nervous system disorders) | 1 | 3
Convulsion (Nervous system disorders) | 5 | 2
Irritability (Psychiatric disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days